CLINICAL TRIAL: NCT02362945
Title: Hexakaprone Treatment for Post-Partum Hemorrhage Prophylactic
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yariv yogev (Other)
Collaborators: Rabin Medical Center (Other)
Responsible Party: Sponsor-Investigator, Yariv yogev, Prof. Yariv Yogev Director, Division of obstetrics and delivery, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0656-14
Record Dates: First submitted 2015-01-15; First posted 2015-02-13 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Post-Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group: (Experimental): Treatment with 1 gr hexakapron Intra-Venous (IV) after delivery of the fetus in addition to accepted treatment with oxytocin (10 units in 100ml NaCl (sodium chloride)0.9% solution IV). ( the oxytocin is the routine practice in our department).
  Interventions: Drug: Intervention group:
- Control: (No Intervention): Treatment with oxytocin after fetal extraction (10 units in 100ml NaCl 0.9% solution IV). as commonly given for Post-Partum Hemorrhage (PPH) at our obstetrical ward.Active Comparator: (this is the routine practice in our department).

INTERVENTIONS:
Drug: Intervention group: — Treatment with 1 gr hexakapron Intra-Venous (IV) after delivery of the fetus in addition to accepted treatment with oxytocin (10 units in 100ml NaCl 0.9% solution IV).
  Other Names: Hexakaprone-Transexamic acid and oxytocin
  Arms: Intervention group:

SUMMARY:
Post-Partum Hemorrhage (PPH) is a common obstetrical complication. It may occur after both vaginal and cesarean delivery with a reported prevalence of 4-6% of deliveries [1]. Prophylactic treatment with oxytocin after fetus extraction is a common practice. [1,2]Transexamic acid - Hexakapron is a potent antifibrinolytic, it prevents lysine adhesion to plasminogen molecules by blocking its binding site. It can lower fibrinolysis rate and by that reduce bleeding [9]. Systematic treatment of anti-fibrinolytic drugs is in surgical practice after procedures such as coronary artery bypass graft, orthopedic surgeries and liver transplantation [10-13]. Hexakapron is an FDA approved drug, it is defined as a class B drug for pregnancy and lactation [12], it is already being used in a non-routine fashion in the delivery room during PPH.In obstetrics Hexakapron given before vaginal or cesarean delivery has been presumed to decrease blood loss and PPH. 2 studies that included 453 woman reported decrease in PPH (RR 0.51, 95% CI 0.36 to 0.72) [13-15]. However specific protocols for prophylactic treatment with Hexakapron as available with oxytocin are lacking, and further research is necessary to determine such guidelines [16].

DETAILED DESCRIPTION:
Post-Partum Hemorrhage (PPH) is a common obstetrical complication. It may occur after both vaginal and cesarean delivery with a reported prevalence of 4-6% of deliveries [1]. Prophylactic treatment with oxytocin after fetus extraction is a common practice. [1,2] The increase in plasma volume during pregnancy, and uterine perfusion that reaches 750ml/min near term [3] are causes for excessive blood loss during vaginal or cesarean delivery. Blood loss is approximately 500ml and 1000ml during vaginal and cesarean delivery respectively. Studies have shown that blood transfusion treatment reaches to up to 6 % after cesarean section [5-6].

During placental delivery fibrinogen and fibrin degradation and plasminogen activation occurs. This causes fibrinolytic cascade that continues 6-10 hours post-partum [7]. Tissue injury during cesarean section may convert the hemostatic equilibrium towards fibrinolysis that results in excessive bleeding [8]/ Transexamic acid - Hexakapron is a potent antifibrinolytic, it prevents lysine adhesion to plasminogen molecules by blocking its binding site. It can lower fibrinolysis rate and by that reduce bleeding [9]. Systematic treatment of anti-fibrinolytic drugs is in surgical practice after procedures such as coronary artery bypass graft, orthopedic surgeries and liver transplantation [10-13]. Hexakapron is an FDA approved drug, it is defined as a class B drug for pregnancy and lactation [12], it is already being used in a non-routine fashion in the delivery room during PPH.

In obstetrics Hexakapron given before vaginal or cesarean delivery has been presumed to decrease blood loss and PPH. 2 studies that included 453 woman reported decrease in PPH (RR 0.51, 95% CI 0.36 to 0.72) [13-15]. However specific protocols for prophylactic treatment with Hexakapron as available with oxytocin are lacking, and further research is necessary to determine such guidelines [16].

PPH jeopardize young reproductive women's health, it is specifically related to major morbidity in the context of prior anemia which features this population in high rates [17]. PPH is the major maternal cause of death, with 100000 cases per year [6].

Thus the investigators sought to investigate the efficacy of Hexakapron, as a prophylactic treatment after vaginal delivery and cesarean section, in reducing PPH.

ELIGIBILITY:
Inclusion Criteria:

* Normal vaginal delivery.
* Operative vaginal delivery (Vaccum and Forceps).
* Elective cesarean section.
* Age 18-50.

Exclusion Criteria:

* Excessive pain (VAS>4).
* Blood clotting disturbance or any major hematologic disease.
* Suspected Placenta-Previa.
* Multiple gestations.
* Contraindications for Hexakapron treatment:

  * Atrial fibrillation.
  * Coronary arteries stenting.
  * CABG(coronary artery bypass graft) in past year.
  * Hematuria (prior to pregnancy).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Decrease post-partum hemoglobin decline. | 24 month
  Assessment of the hemoglobin decline - the decline will be calculated as the gap between the hemoglobin level prior delivery and the the hemoglobin measured 48-72 hours post delivery.

SECONDARY OUTCOMES:
Decrease PPH. | 24 month
  rates of Post-partum hemorrhage will be assessed by The difference between the groups
Decrease the need for post-partum uterine manual revision. | 24 month
  rates of Post-partum uterine manual revision will be assessed by The difference between the groups the difference will be assessed by a chi-square test.

CONTACTS AND LOCATIONS:
Overall Officials: Yariv Yogev, professor, Principal Investigator — Director, Division of obstetrics and delivery